CLINICAL TRIAL: NCT04801082
Title: Endoscopic Ultrasound-Guided Coeliac Plexus Neurolysis for Cancer Pain: Chemical Versus Radiofrequency Ablation
Brief Title: Endoscopic Ultrasound Guided Coeliac Plexus Neurolysis for Cancer Pain
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Ma Ka Wing, Clinical Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202009185043
Record Dates: First submitted 2021-03-08; First posted 2021-03-16 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Malignancy; Pain Management
Keywords: Endoscopic Ultrasound Guided; Radiofrequency Ablation; Coeliac plexus neurolysis; Intra-abdominal malignancy; Pain Relief; Chemical coeliac plexus neurolysis; Coeliac plexus ablation; Cancer pain
MeSH Terms: conditions — Neoplasms; Agnosia; Cancer Pain | interventions — Ethanol; Radiofrequency Ablation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- EUS-CPB (Active Comparator): Endoscopic Ultrasound Guided Coeliac Plexus Block
  Interventions: Drug: Alcohol injection
- EUS-CPA (Active Comparator): Endoscopic Ultrasound Guided Coeliac Plexus Radiofrequency Ablation
  Interventions: Device: Radiofrequency Ablation

INTERVENTIONS:
Drug: Alcohol injection — Chemical ablation is performed by injection of 10 mL of 0.25% bupivacaine, followed by 10 mL of 98% dehydrated alcohol using a 22G FNA needle (Cook and Olympus)
  Other Names: Chemical Ablation
  Arms: EUS-CPB
Device: Radiofrequency Ablation — coeliac plexus is identified and punctured with 19G EUSRA RFA needle with 10W-30W of energy for 10-50s bilaterally or unilaterally depends on individual anatomical characteristics.
  Other Names: RFA
  Arms: EUS-CPA

SUMMARY:
Many cancer patients suffer from intractable pain and which is often suboptimally controlled by even strong opioid analgesics. Coeliac plexus neurolysis (CPN) is procedure which intended to permanently destroy the nociceptive pathway that transmits the pain caused by the tumour. It can be with different approaches, such as percutaneously guided by fluoroscopy, echo-endoscopically or surgically with endoscopic approach being the more popular one in many centers equipped with echo-endoscopic services. The effect of CPN has been well established by some retrospective series. The overall response rate to CPN ranges from 70-90%, however, the analgesic effect is limited and up to roughly around 3 months. It is believed that the short-lasting analgesic effect is related to incomplete neurolysis by absolute alcohol injection.

Recently, radiofrequency ablation (RFA) of coeliac plexus has been introduced as another mode of CPN. So far, only one small single center randomized controlled trial (RCT) suggesting superior performance in favour to CPN using RFA. This result has to be validated and by a RCT with larger sample size. In addition, data concerning the quality of life (QOL) improvement and cost-effectiveness need to be further elucidated. Therefore, the aim of this study is to perform a RCT to look into these issues.

DETAILED DESCRIPTION:
The aim of this study is to compare the efficacy of EUS-CPN by chemical ablation using alcohol injection versus by radiofrequency ablation in patients with cancer pain related to intra-abdominal malignancy. This is a randomised controlled trial to assess the clinical outcomes and cost-effectiveness of this new treatment approach.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 year-old
* Patients who give informed consent to the study
* Suboptimal pain control with regular analgesics
* Inoperable cancer of pancreas, biliary system and liver (both primary or secondary)

Exclusion Criteria:

* Patients who refuse to give consent
* Patients aged <18 years
* EUS not possible due to:
* Problem related to scope insertion such as trismus, stenosis of the upper GI tract
* Coagulopathy with INR >1.5 or platelet count < 70
* Low oxygen saturation or extreme blood pressure render endoscopic procedure unsafe

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2024-01-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Change of pain score | 4 weeks after the procedure
  change of pain score at 4th week after the procedure (by VAS score)

SECONDARY OUTCOMES:
Change of pain score | 2 weeks, 4 weeks, 8 weeks, 12 weeks, 24 weeks
  change of pain score (Visual Analog Score) after the procedure
Analgesic requirement | Up to 100 months (From the date of procedure until the date of death from any cause)
  decrease in analgesic requirement
Technical success rate | 1 day
  technical success rate
Clinical success rate | Through study completion, an average of 2 year
  decrease in pain level by 30% from the pre-procedural baseline
Duration of procedure | Up to 1 hour
  time from injection of pre-medication to procedure last observation recording at the procedure suite
Time to pain score drop by 50% | Through study completion, an average of 2 year
  Time to Visual Analog Score drop by 50%
Short term complication rate | Up to 1 week
  complication rate
Long term complication rate | Through study completion, an average of 2 year
  complication rate
Hospital length of stay | Up to 100 months
  Hospital length of stay
Health status (Quality of life) | 2 weeks, 4 weeks, 8 weeks, 12 weeks, 24 weeks
  The Short Form (36) Health Survey
Quality of life (QOL) in patients with pancreatic cancer | 2 weeks, 4 weeks, 8 weeks, 12 weeks, 24 weeks
  PAN-26 questionnaire
Quality of life (QOL) of cancer patients | 2 weeks, 4 weeks, 8 weeks, 12 weeks, 24 weeks
  QLQ-C30 questionnaire
Cost-effectiveness | Through study completion, an average of 2 year
  Total cost ($) of the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ka Wing Ma, MBBS, MS, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong